CLINICAL TRIAL: NCT02303119
Title: A Randomized Phase III Trial Evaluating Two Strategies of Rituximab Administration for the Treatment of First Line/Low Tumor Burden Follicular Lymphoma (Follicular Lymphoma IV/SC Rituximab Therapy)
Brief Title: Follicular Lymphoma IV/SC Rituximab Therapy (FLIRT)
Acronym: FLIRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLIRT
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Follicular Lymphoma
Keywords: LNH; CD20+; follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Am A : Rituximab IV (Active Comparator): 4 infusions of intravenous rituximab (375mg/m²) at Day 1, Day 8, Day 15 and D22
  Interventions: Drug: Rituximab IV
- Arm B: Rituximab SC (Experimental): 1 infusion of intravenous rituximab (375mg/m²) at Day 1, and 7 administrations of sub-cutaneous rituximab (1400mg) at Day 8, Day15, Day 22, Month 3, Month 5, Month 7 and Month 9.
  Interventions: Drug: Rituximab IV; Drug: Rituximab SC
- Arm C : Rituximab SC first cycle (Experimental): 8 administrations of sub-cutaneous rituximab (1400mg) at Day 8, Day15, Day 22, Month 3, Month 5, Month 7 and Month 9.
  Interventions: Drug: Rituximab SC

INTERVENTIONS:
Drug: Rituximab IV — intra-venous, 375 mg/m²
  Other Names: MabThera IV
  Arms: Am A : Rituximab IV; Arm B: Rituximab SC
Drug: Rituximab SC — sub-cutaneous, 1400 mg
  Other Names: MabThera SC
  Arms: Arm B: Rituximab SC; Arm C : Rituximab SC first cycle

SUMMARY:
Patient will receive either one infusion of rituximab IV and seven administrations of rituximab SC (experimental arm) or four infusions of rituximab IV (standard arm).

The hypothesis is that the use of rituximab by sub cutaneous route and the scheme of administration could:

* optimize rituximab exposure leading to improve response rate
* increase adaptative response and then improve long-term control disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma CD20+ grade 1, 2 and 3a by biopsy within 4 months before signing informed consent
* Have a bone marrow biopsy within 4 months before the first study drug administration
* Have no prior therapy except surgery for diagnosis
* Aged 18 years or more with no upper age limit
* ECOG performance status 0-2
* Ann Arbor Stage II, III or IV
* Bi-dimensionally measurable disease defined by at least one single node or tumor lesion > 1.5 cm assessed by CT scan and/or clinical examination
* With low-tumor burden defined as:

  * Nodal or extra-nodal tumor mass with diameter less than 7 cm in its greater diameter
  * And involvement of less than 3 nodal or extra nodal sites with diameter greater than 3 cm
  * And absence of B symptoms
  * And no symptomatic splenomegaly
  * And no compression syndrome (ureteral, orbital, gastrointestinal…)
  * And no pleural or peritoneal serous effusion
  * And no cytopenia, with hemoglobin > 10 g/dL (6.25mmol/L) and absolute neutrophil count> 1.5 G/L and platelets > 100 G/L within 28 days before the randomization
  * And LDH < ULN within 28 days before the randomization
  * And β2 microglobulin < ULN within 28 days before the randomization
* Have signed an informed consent
* Must be covered by a social security system

Exclusion Criteria:

* Grade 3b follicular lymphoma
* Ann Arbor Stage I
* Seropositive for or active viral infection with hepatitis B virus (HBV) HBs Ag positive HBs Ag negative, anti-HBs antibody positive and/or anti-HBc antibody positive and detectable viral DNA

Note:

Patients who are HBs Ag negative, anti-HBs positive and/or anti-HBc positive but viral DNA negative are eligible Patients who are seropositive due to a history of hepatitis B vaccine are eligible

* Known seropositive for, or active viral infection with hepatitis C virus (HCV)
* Known seropositive for, or active viral infection with Human Immunodeficiency Virus (HIV)
* Any of the following laboratory abnormalities within 28 days before the randomization:

Total bilirubin or GGT or AST or ALT > 3 ULN. Calculated creatinine clearance (Cockcroft and Gault formula) < 60 mL /min

* Presence or history of CNS involvement by lymphoma
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patient with mental deficiency preventing proper understanding of the informed consent and the requirements of treatment.
* Adult under law-control
* Adult under tutelage
* Contraindication to use rituximab or known sensitivity or allergy to murine products
* Pregnant or lactating females.
* Concomitant disease requiring prolonged use of corticosteroids or corticosteroids administration for lymphoma within 28 days before the first study drug administration.
* Male and female patients of childbearing potential who cannot or do not wish to use an effective method of contraception, during the study treatment and for 12 months thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5.5 years
  Time from randomization into the study to the first observation of documented disease progression or death due to any cause. If a subject has not progressed or died, PFS will be censored at the time of last visit with adequate assessment

SECONDARY OUTCOMES:
Overall Survival (OS) | 5.5 years
  time from the date of randomization to the date of death from any cause. Alive patients will be censored at their last follow-up date.
Response Rates | M3 and M12
  Disease response evaluation, assessment will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma) according to Cheson 1999 (M3 and M12) and according to Cheson 2014 (M12 only).
  The response rates will be described for each modality (CR, CRu, PR, SD and PD) and the Overall response rates (CR+CRu+PR) will also be described at the two time points (M3 & M12).
Best Response Rate during the study | M3 and M12
  Best disease response, assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999)).
  The response rates will be described for each modality (CR, CRu, PR, SD and PD) and the Overall response rates (CR+CRu+PR) will also be described
Time to Next Anti-Lymphoma Treatment (TTNLT) | 5.5 years
  time from randomization to the date of first documented administration of any new anti-lymphoma treatment (chemotherapy, radiotherapy, radio-immunotherapy, immunotherapy…). Patients continuing in response or who are lost to follow-up will be censored on their last visit date. Patients who died (due to any cause) before having received a new anti-lymphoma treatment will be included in the statistical analysis with death being counted as an event.
Molecular Response | M3 and M12
  Bcl-2-IgH rearrangement

OTHER OUTCOMES:
Pharmacokinetic parameters of rituximab will be used to estimate individual area under the concentration curves of rituximab (AUC). | 5.5 years
  The AUC will be used to describe the relationship between rituximab pharmacokinetics and clinical response (objective response, survival).
Causes of death | 5.5 years
  classification by cause of death
Secondary cancers | 5.5 years
  classification by type of cancer
Number of SAE from the first administration | 1 year
  for Rituximab SC as of C1 cohort

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Cartron, MD PhD, Study Chair — Lymphoma Study Association
Locations (50):
- France (50):
  - CH de Pays d'Aix, Aix-en-Provence
  - CHU Angers, Angers
  - CH d'Avignon - Hôpital Henri Duffaut, Avignon
  - Hôpital de Bayonnes, Bayonne
  - CH de BLOIS, Blois
  - Hôpital d'Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - IHBN - CHU de Caen, Caen
  - Clinique du Parc, Castelnau-le-Lez
  - CH de Chambéry, Chambéry
  - Chu Estaing, Clermont-Ferrand
  - Hôpital Pasteur, Colmar
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon - Hôpital d'Enfants, Dijon
  - Hôpital Albert Michallon, Grenoble
  - CH Départemental Vendée, La Roche-sur-Yon
  - Hôpital St Louis, La Rochelle
  - Hôpital André Mignot, Le Chesnay
  - Clinique Victor Hugo, Le Mans
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Conception, Marseille
  - Hôpital Mercy, Metz
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Institut de Cancérologie du Gard Hématologie clinique, Nîmes
  - CHR de la Source, Orléans
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint Jean, Perpignan
  - Hôpital Haut Lévêque - Centre François Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CH René Dubos, Pontoise
  - Centre Hospitalier Annecy-Genevois, Pringy
  - Hôpital Robert Debré, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Victor Provo, Roubaix
  - Centre Henri Becquerel, Rouen
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital de Hautepierre, Strasbourg
  - IUCT Oncopole, Toulouse
  - Hôpital Bretonneau, Tours
  - CH de TROYES, Troyes
  - CH de Valenciennes, Valenciennes
  - CHU Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cartron G, Bachy E, Tilly H, Daguindau N, Pica GM, Bijou F, Mounier C, Clavert A, Damaj GL, Slama B, Casasnovas O, Houot R, Bouabdallah K, Sibon D, Fitoussi O, Morineau N, Herbaux C, Gastinne T, Fornecker LM, Haioun C, Launay V, Araujo C, Benbrahim O, Sanhes L, Gressin R, Gonzalez H, Morschhauser F, Ternant D, Xerri L, Tarte K, Pranger D. Randomized Phase III Trial Evaluating Subcutaneous Rituximab for the First-Line Treatment of Low-Tumor Burden Follicular Lymphoma: Results of a LYSA Study. J Clin Oncol. 2023 Jul 1;41(19):3523-3533. doi: 10.1200/JCO.22.02327. Epub 2023 Apr 18. PMID 37071836